CLINICAL TRIAL: NCT06225206
Title: Retrospective Exploratory Analysis of Donor-derived Cell Free DNA in Liver Transplant Patients
Brief Title: Analysis of Donor-derived Cell Free DNA in Liver Transplant Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 023.HEP.2023.D
Record Dates: First submitted 2023-11-13; First posted 2024-01-25 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-01

CONDITIONS: Liver Transplant Failure
MeSH Terms: interventions — Liver Extracts

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: donor-derived cell free DNA in liver — Determine the difference in age, gender, LFTs, IS regimen (tacrolimus/sirolimus/cyclosporin with mycophenolate mofetil (MMF) and /or prednisone) between patients who underwent liver transplant <1 year PTX and >1 year PTX

SUMMARY:
Determine the levels of Donor-derived (dd)cell-free DNA(cfDNA )in liver transplant recipients with normal liver function tests (LFTs) indicating stable immunosuppression status (IS). Based on this range use the dd-cfDNA levels to determine over or under IS in liver transplant patients to make changes to their IS medication regimen.

DETAILED DESCRIPTION:
dd-cfDNA is a non-invasive method to measure graft function stability in liver transplant patients. Liver biopsy is the standard to determine liver rejection and graft function, but no tests exist currently to be able to help guide the IS regimen in these patients. LFTs are not as specific to determine graft function hence testing dd-cfDNA levels can help guide the Immunosuppression (IS )medications dosing and help identify rejection early.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years
2. The patient underwent a liver transplant.
3. The patient at least has one level of dd-cfDNA documented

Exclusion Criteria:

* Patient not meeting the inclusion criteria will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the study should be at least 18 years of age, who have underwent a liver transplant and at least have one level of dd-cfDNA documented.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
dd-cfDNA range in liver transplant patients | 1 year
  Determine the dd-cfDNA in liver transplant patients with stable IS collected from July 2021 to July 2024 and compare the range between patients with <1-year post-transplant (PTX) and >1-year PTX by chart review using Methodist hospital data system.

SECONDARY OUTCOMES:
Demographics: age (years), gender (male/female), race (Caucasian, Black, Hispanic, Asian, Other) | 1 year
  Demographics differences in patients who underwent liver transplant less than 1 year of PTX and more than 1 year PTX
Days post-transplant at first dd-cfDNA | 1 year
  Number of days post transplant at first dd-cfDNA
LFTs: Alanine transaminase(ALT), Aspartate transaminase(AST),Alkaline phosphatase( ALP), total bilirubin (Tbili) | 1 year
  looking at the liver function tests in patients who underwent liver transplant less than 1 year of PTX and more than 1 year PTX
Serum Creatinine | 1 year
  Measuring the serum creatinine levels

CONTACTS AND LOCATIONS:
Overall Officials: Parvez Mantry, MD, Principal Investigator — Methodist Midlothian Medical Center
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data or any protected health information will not be shared with anyone that is not delegated to the study. The PI is committed to disseminate research results in a timely fashion. Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals
Time Frame: 2 years